CLINICAL TRIAL: NCT02753374
Title: Registry Study on Cystic Fibrosis in Chinese Children-a Multicenter, Prospective Cohort Study
Brief Title: Registry Study on Cystic Fibrosis in Chinese Children
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Children's Hospital (Other)
Collaborators: Shengjing Hospital (Other); Capital Institute of Pediatrics, China (Other); Shanghai Children's Medical Center (Other); Shenzhen Children's Hospital (Other Government); The First Affiliated Hospital of Xiamen University (Other); First Affiliated Hospital of Guangxi Medical University (Other)
Responsible Party: Principal Investigator, Kunling Shen, Chief of China National Clinical Research Center for Respiratory Diseases, Beijing Children's Hospital
Other Study IDs: BCHlung004
Record Dates: First submitted 2016-04-26; First posted 2016-04-27 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis, Chinese, children
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study is a multicenter, prospective cohort study of patients diagnosed with cystic fibrosis, the clinical information of recruited patients, including clinical manifestations, lung function, chest imaging, quality of life and other indicators, will be followed for 10 years.

DETAILED DESCRIPTION:
All new cases of cystic fibrosis which was confirmed or probably diagnosed at each center from the beginning of the study are made the investigation of the clinical manifestations, sweat test and CFTR mutations by the standard diagnostic process.Then all the patients' following clinical data will be followed for 10 years (once per six month): clinical manifestations, lung function, chest imaging (once per year), quality of life and other indicators.

ELIGIBILITY:
Inclusion Criteria:

* Age 0~18 years old
* Any organ system symptoms consistent with CF, such as chronic sinopulmonary disease, gastrointestinal and nutritional abnormalities, obstructive azoospermia or having siblings with CF
* CFTR dysfunction indicated by elevated sweat chloride levels ≥60 mmol/L twice, or one sweat chloride levels ≥40 mmol/L plus presence of two pathogenic CFTR mutations on different alleles
* Probable CF patients with sweat chloride levels among 40~59 mmol/L plus with presence of 0-1 pathogenic CFTR mutation
* Consent to provide the related clinical specimen to the certain hospital
* The guardians of the patients fully understand the purpose of the study, volunteer their children to participate in this study and sign informed consent.

Exclusion Criteria:

* Subject will be excluded if she or he has one of the following:
* It is unable to provide complete medical records or the current condition can not accept the diagnosis process.
* She or he does not agree to participate in the test.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children who was confirmed diagnosis as cystic fibrosis at the certain hospitals (sponsor and collaborators)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-05; Primary Completion 2030-05 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in lung function on the spirometry | ten years
  forced expiratory volume at one second (FEV1) in Liter

CONTACTS AND LOCATIONS:
Overall Officials: Kunling Shen, MD, PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China, China National Clinical Research Center for Respiratory Diseases; Baoping Xu, MD, PhD, Principal Investigator — Beijing Children's Hospital of Capital Medical University, China, China National Clinical Research Center for Respiratory Diseases

REFERENCES:
- [Background] Kerem B, Rommens JM, Buchanan JA, Markiewicz D, Cox TK, Chakravarti A, Buchwald M, Tsui LC. Identification of the cystic fibrosis gene: genetic analysis. Science. 1989 Sep 8;245(4922):1073-80. doi: 10.1126/science.2570460.
- [Background] Comeau AM, Parad RB, Dorkin HL, Dovey M, Gerstle R, Haver K, Lapey A, O'Sullivan BP, Waltz DA, Zwerdling RG, Eaton RB. Population-based newborn screening for genetic disorders when multiple mutation DNA testing is incorporated: a cystic fibrosis newborn screening model demonstrating increased sensitivity but more carrier detections. Pediatrics. 2004 Jun;113(6):1573-81. doi: 10.1542/peds.113.6.1573. PMID 15173476
- [Background] Nazer HM. Early diagnosis of cystic fibrosis in Jordanian children. J Trop Pediatr. 1992 Jun;38(3):113-5. doi: 10.1093/tropej/38.3.113. PMID 1507302
- [Background] Al-Mahroos F. Cystic fibrosis in bahrain incidence, phenotype, and outcome. J Trop Pediatr. 1998 Feb;44(1):35-9. doi: 10.1093/tropej/44.1.35. PMID 9538604
- [Background] Yamashiro Y, Shimizu T, Oguchi S, Shioya T, Nagata S, Ohtsuka Y. The estimated incidence of cystic fibrosis in Japan. J Pediatr Gastroenterol Nutr. 1997 May;24(5):544-7. doi: 10.1097/00005176-199705000-00010. PMID 9161949
- [Background] Brennan ML, Schrijver I. Cystic Fibrosis: A Review of Associated Phenotypes, Use of Molecular Diagnostic Approaches, Genetic Characteristics, Progress, and Dilemmas. J Mol Diagn. 2016 Jan;18(1):3-14. doi: 10.1016/j.jmoldx.2015.06.010. Epub 2015 Nov 26. PMID 26631874